CLINICAL TRIAL: NCT01415258
Title: Screening for Vulnerability in the Elderly Supported at the Oscar Lambret Centre
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Hôpital Gériatrique Les Bateliers, CHRU Lille (Unknown)
Responsible Party: Sponsor
Other Study IDs: VULNERABILITE-1103
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Solid Tumor
Keywords: cancer; vulnerability; frail
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to uncover the prevalence of vulnerability among patients aged ≥ 70 coming to the medical oncology division of the Oscar Lambret Centre, according to the short screening test Vulnerable Elders Survey 13 (VES-13).

The objective is to better understand the value of routine screening of patients before the consultation, it was proposed as a secondary objective of this study to assess the correlation between the identification of the vulnerability in the screening test VES-13 and the identification made by the clinician during the consultation. The correlation between VES-13 and opinion of the clinician for three categories of patients (self - intermediate - fragile) will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* patient aged ≥ 70
* coming for a first visit, whatever the purpose and the disease stage

Exclusion Criteria:

* neglect or refusal to answer to the VES-13 test

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study concerns elderly patients (≥70 years) with solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To assess the Vulnerable Elders Survey score (VES-13) | Within 3 months after recruitment
  A patient is identified vulnerable if the score is ≥ 3

SECONDARY OUTCOMES:
To assess the correlation between the VES-13 score and the vulnerability judged by a clinical expert | Within 3 months after recruitment
  A patient will be identified as vulnerable if he/she belongs to the "intermediate" or "frail" category. The Kappa coefficient of agreement will be used to correlate the VES-13 score and clinical observations.
To measure the muscle strength using the grip strength test | Within 3 months after recruitment
  Hand Dynamometer Range values : 0-90

CONTACTS AND LOCATIONS:
Overall Officials: Véronique SERVENT, MD, Principal Investigator — Oscar Lambret Anti-Cancer Centre
Locations (1):
- Oscar Lambret Anti-Cancer Centre, Lille, France